CLINICAL TRIAL: NCT03663595
Title: Effects of Two Treatment Models on Neuromuscular Properties of Young Women Symptomatic for Patellofemoral Pain Syndrome: A Randomized Controlled Trial
Brief Title: Treatment Effects on Neuromuscular Properties on Young Women Symptomatic for Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Marco Aurélio Vaz, PhD, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UFRGS - 2.809.328
Record Dates: First submitted 2018-08-30; First posted 2018-09-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral pain; Etiology; Multiarticular rehabilitation; Local factors; Nonlocal factors
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PFPS: Model 1 (Hip and Knee) (Experimental): Females symptomatic for PFPS. This group will be submitted to the rehabilitation program with exercises focusing in proximal (hip) and local (knee) factors.
  Interventions: Other: Model 1
- PFPS: Model 2 (knee, foot and ankle) (Experimental): Females symptomatic for PFPS This group will be submitted to the rehabilitation program with exercises focusing in distal (foot and ankle) and local (knee) factors.
  Interventions: Other: Model 2
- Healthy group (No Intervention): Healthy females not submitted to intervention

INTERVENTIONS:
Other: Model 1 — Model 1 will be composed of exercises focusing on local (knee) and proximal (hip) factors.
  Other Names: Local and proximal factors
  Arms: PFPS: Model 1 (Hip and Knee)
Other: Model 2 — Model 2 will be composed of exercises focused on the local (knee) and distal (ankle and foot) factors.
  Other Names: Local and distal factors
  Arms: PFPS: Model 2 (knee, foot and ankle)

SUMMARY:
Patellofemoral Pain Syndrome (PFPS) is characterized by diffuse pain around the knee joint. This presence of pain is the most common manifestation in sports medicine among adults and young people. Women are more likely to develop PFPS. Among the young adult population, it is estimated that 13% of the women are affected by PFPS. There is a consensus among clinicians that PFPS etiology is multifactorial, including local factors (structures present or acting directly on the patellofemoral joint) and nonlocal factors [extrinsic to the patellofemoral joint, including proximal factors (hip, trunk and pelvis), and distal factors (ankle and foot)]. PFPS is not a degenerative syndrome, and conservative treatment offers good results. However, the most appropriate therapeutic approach is still unclear, and the rate of nonresponders to treatment is high. One of the possible explanations for failure of the therapeutic intervention is that the triggering mechanisms of PFPS are not the same for all subjects, and probably some patients cannot be reached by standard treatment. The traditional intervention model focuses on the strengthening of the knee extensor muscles, but recent literature has pointed out that multi-articular treatment models (i.e., exercises for the proximal or distal factors, in addition to exercises for the quadriceps) have shown better results. It is believed that the elaboration of treatment protocols combining local and non-local factors, present greater responsiveness and results retention, thus reducing treatment failure. Based on this, and due to the lack of experimental studies that aimed to compare the effects of a multi-articular intervention protocol combining local and non-local factors in women affected by PFPS, this study aims to evaluate the effects of two multi-articular intervention protocols based on exercises (1) for the proximal and local factors versus (2) for the distal and local factors on the clinical, functional and neuromechanical outcomes of young women with PFPS. Participants of the PFPS group will be submitted to one of two intervention models for an 12-week rehabilitation program. Model 1 will be composed of exercises focusing on local and proximal PFPS factors, and Model 2 will be composed of exercises focused on the local and distal factors.

DETAILED DESCRIPTION:
Healthy females (CG, n=20) were not submited to intervention and PFP participants will be divided into 2 intervention groups (PFPS group, n=66). PFPS Participants' inclusion in the study will be done based on their anamnesis and clinical tests. Participants will be recruited primarily at the School of Physical Education, Physical Therapy and Dance of the Federal University of Rio Grande do Sul (UFRGS). The PFPS group will be submitted to one of two intervention models based on physical exercises, with an 12-week duration, and 2 sessions per week. Model 1 will be composed of exercises focusing on local and proximal factors, and Model 2 will be composed of exercises focused on the PFPS local and distal factors. Only the PFPS group will receive the intervention program. The allocation of each participant's intervention model will be randomized. All participants will be submitted to the following evaluations: (1) anthropometric measurements (mass, height and body mass index), (2) self reported functionality (Kujala Questionnaire), (3) single leg squat and drop landing tests (kinematic analysis), (4) muscle strength (evaluated with a hand held dynamometer), (5) pain (evaluated by numeric pain rating scale), (6) muscle activation (evaluated by EMG) and (7) muscle thickness (evaluated by ultrasonography).

ELIGIBILITY:
Patellofemoral pain syndrome group:

Inclusion Criteria:

A physiotherapist evaluated PFP participants' eligibility based on the following criteria: (1) presence of peripatelar or retropatelar pain in at least two functional tasks (squatting, running, kneeling, jumping, climbing or descending stairs, sitting for a long time, sitting with knees flexed), (2) ongoing patellar pain for at least 3 months, (3) PFP with a minimum of 3 out of 10 points in the numeric rating scale for knee pain (0 = "no pain", 10 = "intolerable pain"), (4) beginning of PFP symptoms not related to trauma and (5) not participating in any PFP treatment in the last 12 months

Exclusion Criteria:

* Participants were excluded if they presented signs or symptoms of (1) meniscal or other intra-articular pathologies; (2) signs of patellar apprehension; (3) history of hip, knee, or ankle joint injury; (4) evidence of joint effusion; and (5) history of patellofemoral joint surgery.

Healthy group (n=20): women with no history of PFP in the last 12 months

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change of knee pain | The evaluation will be performed to baseline (pre-intervention), change from baseline to 6 weeks of intervention and change from baseline to 12 weeks of intervention.
  Knee pain will be measured with a Numeric Pain Rating Scale (0 to 10)
Self-reported functionality | The evaluation will be performed to baseline (pre-intervention), change from baseline to 6 weeks of intervention and change from baseline to 12 weeks of intervention.
  Self-reported functionality will be measured by Anterior Knee Pain Scale by Kujala Questionaire (1993)
Change in knee muscles, hip muscles, ankle muscles and foot muscles strength | The evaluation will be performed to baseline (pre-intervention), change from baseline to 6 weeks of intervention and change from baseline to 12 weeks of intervention.
  Torque is an expression of the muscular strength and was assessed by dynamometry
Change of kinematic of pelvis, hip, knee and ankle during single leg squat | The evaluation will be performed to baseline (pre-intervention), change from baseline to 6 weeks of intervention and change from baseline to 12 weeks of intervention.
  Single leg squat will be measured with a video camera, and will be used to determine lower limb alignement
Change of kinematic of pelvis, hip, knee and ankle during drop landing test | The evaluation will be performed to baseline (pre-intervention), change from baseline to 6 weeks of intervention and change from baseline to 12 weeks of intervention.
  rop landing will be measured with a video camera, and will be used to determine lower limb alignement
Change of knee muscles, hip muscles, ankle muscles and foot muscles architecture | The evaluation will be performed to baseline (pre-intervention), change from baseline to 6 weeks of intervention and change from baseline to 12 weeks of intervention.
  Muscular architecture (muscle thickness) will be assessed by ultrasonography
Muscle activation | The evaluation will be performed to baseline (pre-intervention), change from baseline to 6 weeks of intervention and change from baseline to 12 weeks of intervention.
  Muscle activation will be assessed by electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Marco Vaz, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Exercise Research Laboratory, School of Physical Education, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pompeo KD, da Rocha ES, Melo MA, de Oliveira NT, Oliveira DF, Sonda FC, Dos Santos PF, Rodrigues R, Baroni BM, Vaz MA. Can we replace exercises targeted on core/hip muscles by exercises targeted on leg/foot muscles in women with patellofemoral pain? A randomized controlled trial. Phys Ther Sport. 2022 Nov;58:1-7. doi: 10.1016/j.ptsp.2022.08.004. Epub 2022 Aug 28. PMID 36067687